CLINICAL TRIAL: NCT05981716
Title: Factors Affecting Quality of Life and Treatment Adherence Among Early-Age-at-Onset Breast Cancer Survivors
Brief Title: Young Breast Cancer Survivors Study
Acronym: YBCSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Susan Steck, Professor, University of South Carolina
Other Study IDs: YBCSS-2023
Record Dates: First submitted 2023-03-12; First posted 2023-08-08 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Nutrition; Breast Cancer; Cancer Survivors; Quality of Life; Treatment Adherence; Social Determinants
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young Breast Cancer Survivors: The investigators will enroll approximately 384 female breast cancer patients. Only non-institutionalized, English literate, female breast cancer patients diagnosed within the previous ten years and younger than 50 years old at the time of diagnosis will be eligible.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study. There is no intervention.

SUMMARY:
Despite significant overall reductions in mortality rates for breast cancer over the past decade, both incidence and mortality rates have steadily climbed in adults diagnosed before age 50. This research project addresses factors associated with quality of life among and treatment response in early-age-at-onset breast cancer patients. The overall objective is collect information from early-onset breast cancer patients using an online questionnaire and examine factors related to cancer survival, (i.e.,better quality of life, better treatment adherence, less adverse treatment responses).

Aim 1: Identify dietary patterns related to health-related quality of life in early-age-at-onset breast cancer patients. The investigators hypothesize that diet quality is related to better health-related quality of life among young breast cancer survivors.

Aim 2. Identify demographic, social determinants, and geographic factors associated with treatment adherence. The investigators hypothesize that social determinants such as poverty-to-income ratio, education, and proximity to cancer treatment facilities are associated with treatment adherence in early-onset breast cancer.

DETAILED DESCRIPTION:
This is an observational epidemiologic study in which the investigators will collect data from approximately 384 participants at one point in time using online questionnaires (REDCaP and the NCI Diet History Questionnaire III). Recruitment will be conducted via breast cancer survivor social media support groups and advocacy groups. Electronic consent will be granted at the beginning of each online questionnaire. Data collection will occur via self-report in the location chosen by the participant using an online questionnaire. The investigators will use established validated questionnaires used by other previously conducted cohorts to enquire about demographics, occupation, cancer screening history, family history of cancer, comorbidities, cancer and other comorbidity treatment including fertility-related, HRQoL, dietary intake using the online NCI Dietary History Questionnaire III which includes dietary supplement use, residential history, hormonal status, physical activity, tobacco product and alcohol use, experiences with racism, social support, and information on health care utilization.

To accomplish Aim 1, the investigators will use the NCI Diet History Questionnaire III, an online 135-item food frequency questionnaire with 26 dietary supplement questions, reflecting the past one month of intake to estimate food and nutrient intakes and overall dietary patterns.Health related quality of life (HRQoL) is a multidimensional concept that not only includes physical, psychological and social domains, but may also encompass other domains such as cognitive functioning. Cancer patients also exhibit many symptoms (e.g., fatigue, pain, sleep disturbance) that are not measurable directly from laboratory tests. Thus, assessing HRQoL and these symptom burdens among cancer survivors will need to rely on patients' self-reports, measured by validated instruments especially for patients with breast cancer, and includes the Functional Assessment of Cancer Therapy (FACT-B).

Descriptive statistics will be presented as mean (standard deviation) and median (inter quartile range) for continuous variables and as frequency (percentage) for categorical variables. Data visualization tools such as histogram, boxplot, scatterplot and line plot will be employed to assess the trends and outliers in the data. Bivariate association between categorical variables will be tested for statistical significance using Chi-square test or exact test. Differences in continuous variables will be tested for statistical significance using Kruskal-Wallis test. HRQoL data typically are not distributed normally with left-skewed distributions and potential ceiling effects requiring consideration of alternative estimators in multivariate models. A number of different alternative models have been proposed over the standard ordinary least squares approach including beta regression, tobit regression, and two-part modeling. The investigators will assess the distribution of the primary HRQoL measures in building analytic models. With healthy dietary pattern as the primary independent variable and measures of HRQoL serving as primary dependent variable, the investigators expect to find that as diet quality increases, HRQoL increases.

For Aim 2, the investigators will ask study participants to complete questionnaires related to racism, fatalism, and demographics and the investigators will geocode residential histories of participants to measure the role of racism, fatalism, income, education, and proximity to treatment facilities in treatment adherence. The investigators will use geographic information systems to geocode participants' residential histories. Participants will be asked the ZIP code of residence at the time of diagnosis, as well as the ZIP code of the treatment facility in which they received care. If the ZIP code of the treatment facility is unknown, the participant can give the city and state, in which a ZIP code of the central point of the city will be found and used for analysis. Using Microsoft Excel, and the list of latitudes and longitudes by ZIP code, provided by the United States Census Bureau (find citation), the distance in miles between the place of residence and place of treatment will be determined. This distance calculation can be used to help evaluate treatment adherence and the distance to treatment. Residential histories will also be used to determine participant rurality. Regarding the many competing definitions and classification schemes for rurality, Hall et al. found dichotomous definitions mask heterogeneity relevant to health research and studies of accessibility. The investigators will instead use the Rural-Urban Commuting Area (RUCA) codes developed by the Office of Rural Health Policy of the Health Resources and Services Administration and the Economic Research Service of the United States Department of Agriculture (USDA). RUCA codes combine information on population density, urbanicity, and daily commuting patterns to classify census tracts into 22 distinct codes, which can then be consolidated into more manageable classifications.

Descriptive statistics will be presented as mean (standard deviation) and median (inter quartile range) for continuous variables and as frequency (percentage) for categorical variables. Data visualization tools such as histogram, boxplot, scatterplot and line plot will be employed to assess the trends and outliers in the data. The investigators will explore the associations between treatment adherence and each measure of social determinants (such as poverty to income ratio, racism, education, and proximity to treatment facility) using mixed effect logistic regression. The model will be sequentially adjusted for the effect of non-modifiable and modifiable confounders such as age, cancer stage, treatment type, and insurance status.

Recruitment of participants is expected to be ongoing for ~12 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized
* English literate
* Female breast cancer survivors
* Diagnosed with breast cancer within the past 10 years and diagnosed younger than age 50 years

Exclusion Criteria:

* Male breast cancer survivors
* Breast cancer survivors diagnosed with breast cancer after the age of 50 years

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female breast cancer survivors will be considered for the study. There is a much lower prevalence of breast cancer among men; therefore, the study will target a female survivor population.
Study Population: The investigators plan to enroll 384 women who were previously diagnosed with breast cancer prior to the age of 50 years.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Score on Health-related Quality of Life Measure | Measured at one point in time, from 0-10 years after diagnosis
  For Aim 1, health-related quality of life (HRQoL) is a multidimensional concept that not only includes physical, psychological and social domains, but may also encompass other domains such as cognitive functioning. Cancer patients also exhibit many symptoms (e.g., fatigue, pain, sleep disturbance) that are not measurable directly from laboratory tests. Thus, assessing HRQoL and these symptom burdens among cancer survivors will need to rely on patients' self-reports, measured by validated instruments especially for patients with breast cancer. Participants will complete the 37-item Functional Assessment of Cancer Therapy-B with a 5-point Likert-type scale capturing the domains of Physical Well-being, Social/Family Well-being, Emotional Well-being, Functional Well-being, and a Breast Cancer Subscale. Item responses are scored according to scoring guidelines ranging from scores of 0 to 148, with a higher score representing better quality of life.
Number of Participants with Treatment Adherence Compared to those without Treatment Adherence | Up to 2 years post-diagnosis of breast cancer
  For Aim 2, the primary outcome is treatment adherence (at patient-level), which will be determined as per National Comprehensive Cancer Network (NCCN) guidelines and eventually categorized as treatment adherent/non-adherent.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Steck, PhD, MPH, RD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset may be shared with execution of a Data Use Agreement. The study protocol and statistical analysis plan are available upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available at the conclusion of the study after the publication of the main results.
Access Criteria: Contact the Principal Investigator for all requests: Dr. Susan Steck at stecks@mailbox.sc.edu